CLINICAL TRIAL: NCT07226700
Title: A Randomized, Placebo-controlled, Double-blind Trial of Suzetrigine in Total Hip Arthroplasty
Brief Title: Suzetrigine in Total Hip Arthroplasty
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-1169
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Total Hip Arthroplasty (THA); Total Hip Arthroplasty (THA); Total Hip Replacement; Total Hip Replacement Surgery; Total Hip Replacements; Total Hip Replacement Arthroplasty; Suzetrigine; Pain Management; Pain; Nav 1.8; JOURNAVX; Opioid Cessation; Opioid Consumption, Postoperative; Multimodal Analgesia; Randomized Controlled Trial; Randomized Controlled Study; Randomized Controlled Trials
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo arm (Placebo Comparator)
  Interventions: Other: Placebo
- Suzetrigine (Experimental)
  Interventions: Drug: Suzetrigine

INTERVENTIONS:
Drug: Suzetrigine — Suzetrigine is a new novel peripherally acting non-opioid pain medication recently approved by the FDA that exerts its analgesic effects by binding to the peripherally located Nav1.8 Sodium channel receptors present on peripheral nerves.
  Arms: Suzetrigine
Other: Placebo — This will be a placebo drug.
  Arms: Placebo arm

SUMMARY:
Total hip and knee joint replacements are among the most common and painful orthopedic procedures performed worldwide, often requiring intensive analgesia to support early ambulation and recovery. Despite widespread use of multimodal regimens, many patients still rely on opioids, which can cause sedation, nausea, constipation, and long-term dependency. Evaluating Suzetrigine in this high-need population may improve recovery trajectories, reduce opioid consumption, and support enhanced recovery protocols. Given the growing surgical volume and the emphasis on opioid-sparing strategies, rigorous investigation of Suzetrigine's efficacy in joint replacement is of high clinical value. In this study, patients undergoing primary total hip replacement will be randomized to receive either Suzetrigine or placebo for seven days, with the loading dose administered prior to surgery. The primary outcome is cumulative 48-hour opioid consumption in oral morphine equivalents starting from entry into the post-anesthesia care unit (PACU).

DETAILED DESCRIPTION:
Hip and knee replacements are among the most common and painful orthopedic procedures performed worldwide, often requiring intensive analgesia to support early ambulation and recovery. Despite widespread use of multimodal regimens, many patients still rely on opioids, which can cause sedation, nausea, constipation, and long-term dependency. Evaluating Suzetrigine in this high-need population may help inform strategies to improve recovery trajectories, reduce opioid consumption, and support enhanced recovery protocols. Given the growing surgical volume and the emphasis on opioid-sparing strategies, rigorous investigation of Suzetrigine's efficacy in joint arthroplasty is of high clinical value. In this study, patients undergoing primary total hip arthroplasty will be randomized to receive Suzetrigine or placebo for seven days, with the loading dose administered prior to surgery. The primary outcome is cumulative 48-hour opioid consumption in morphine milligram equivalents starting from entry into the post-anesthesia care unit (PACU).

Suzetrigine (VX-548, marketed as Journavx™) is a first-in-class, non-opioid analgesic approved by the U.S. Food and Drug Administration (FDA) in January 2025 for the treatment of moderate-to-severe acute pain in adults [1,2]. It acts through potent and selective inhibition of the voltage-gated sodium channel NaV1.8, which is expressed primarily in peripheral nociceptive neurons (Figure 1) and minimally in the central nervous system [2]. By allosteric stabilization of the channel's closed state (Figure 2), Suzetrigine suppresses nociceptive signaling without impairing cognitive or motor function, offering a novel analgesic mechanism with a low risk of abuse or sedation [3].

Phase III randomized controlled trials have evaluated Suzetrigine for postoperative pain management in procedures such as abdominoplasty and bunionectomy, using the time-weighted sum of the pain intensity difference (SPID) over 48 hours as the primary endpoint [2,4,5]. In these studies, Suzetrigine was compared with placebo and standard opioid regimens. Rescue medications, such as ibuprofen, were permitted.

A supportive phase III safety and effectiveness study (SASE) also assessed Suzetrigine in a broad population that included postoperative surgical and non-surgical patients [6,7]. A subset of these participants underwent orthopedic procedures. In this study, Suzetrigine was administered as a 100 mg loading dose followed by 50 mg every 12 hours for up to 14 days, with acetaminophen and ibuprofen allowed as rescue medications. The most commonly reported adverse events were mild and transient [6,7].

At HSS, multimodal strategies for primary total hip arthroplasty currently include regional anesthesia, acetaminophen, and NSAIDs. Despite these approaches, a proportion of patients still require postoperative opioid prescriptions or refills, suggesting that additional options for acute pain management could be valuable.

Since FDA approval, Suzetrigine has been incorporated into postoperative pain management at HSS for select patients. Evaluating its role in a controlled, randomized setting among patients undergoing THA will provide important data on its use within multimodal protocols and its potential to reduce opioid requirements [5-9].

Suzetrigine, a selective NaV1.8 sodium channel inhibitor, has shown potential for managing acute postoperative pain. However, its clinical utility in broader surgical contexts, such as total hip arthroplasty, remains to be determined. A comprehensive review of the literature and clinicaltrials.gov indicates no randomized controlled trials (RCTs) evaluating Suzetrigine in this population. As such, its efficacy, safety, and opioid-sparing effects in THA have not yet been established.

The primary efficacy outcome used in existing clinical trials evaluating Suzetrigine-specifically in abdominoplasty and bunionectomy procedures-was SPID48 (Summed Pain Intensity Difference over 48 hours). SPID48 is a time-weighted measure based on the Numerical Rating Scale (NRS) for pain collected at multiple time points during the first 48 hours following surgery. While this metric offers a standardized method of assessing pain reduction, further evaluation in large-joint surgery populations is needed to understand its relevance in recovery and functional outcomes.

Additionally, the use of Suzetrigine as a prophylactic perioperative agent-administered before pain onset-has not been explored. This study will address that gap by administering a loading dose prior to surgery. The potential interaction between Suzetrigine and components of contemporary multimodal analgesia, including regional anesthesia and adjunctive medications, also warrants investigation.

No studies to date have evaluated Suzetrigine's effects on subacute pain, functional recovery, or the risk of long-term opioid use. Independent validation is essential to confirm its safety and effectiveness across diverse surgical populations and clinical settings.

In conclusion, while Suzetrigine has been studied in select surgical procedures, its role in managing pain after total hip arthroplasty remains undefined. This study aims to evaluate its efficacy, safety, and opioid-sparing potential in patients undergoing THA and to inform its potential integration into enhanced recovery pathways.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary THA (posterior approach) with participating surgeons
* Age 18 to 80 years old
* Planned discharge to home
* Planned use of neuraxial anesthesia
* American Society of Anesthesiologists (ASA) Physical Status 1 - 3

Exclusion Criteria:

* ASA greater than 3
* Chronic opioid use (daily MME of greater than 30 mg for at least 3 months and within 1 month of surgery)
* History of chronic pain syndromes or uncontrolled pain (i.e. complex regional pain syndrome, fibromyalgia, implanted spinal cord stimulator)
* History of QT prolongation
* Presence of automated implantable cardioverter defibrillator, pacemaker or cardiac resynchronization device
* Evidence of misuse, aberrant use, or addiction to alcohol or an illicitly used drug of abuse, or had a positive test for drugs of abuse
* Inability to comply with any component of the study protocol
* Younger than 18 or greater than 80 years old at the time of enrollment
* Patient already on Suzetrigine
* Allergy or contraindication to Suzetrigine or excipients (eg moderate to severe liver disease/Child Pugh B or C, use of strong CYP3 inhibitors or inducers)
* Contraindications to neuraxial anesthesia or any other part of the study protocol
* Participation in another investigational drug or device study
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-11-03 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption within the first 48 hours after THA starting from PACU entry (t=0), in oral morphine equivalents | From entry into the post-anesthesia care unit (PACU) to 48 hours after THA surgery
  The primary outcome is cumulative 48-hour opioid consumption in oral morphine equivalents starting from entry into the post-anesthesia care unit (PACU). This measure will be taken from EPIC via the MAR and documented in the study "MUD"; post-discharge, patient to report date/time of opioid use # of pills, dose in diary and documented in study "MUD". Measurements will be taken in PACU and 0-48 hrs following surgery.

SECONDARY OUTCOMES:
Post operative pain using Numeric Rating Scale (current at rest, with ambulation, worst & least in last 24 hours) - POD1-7 | From Post Anesthesia Care Unit to post op date 7
  Post operative pain using Numeric Rating Scale (current at rest, with ambulation, worst & least in last 24 hours). The Numeric Rating Scale is a simple, widely used tool for measuring pain intensity. It consists of a 0-10 point scale. This will be measured at post operative day 1 and upto post-operative day 7.
Numeric Rating Scale - PACU: average, least, worst | From arrival in PACU until discharge criteria are met (expected duration up to 4 hours postoperatively).
  Numeric Rating Scale in Post-Anesthesia Care Unit (PACU) ranging from average to least to worst. Post operative pain using Numeric Rating Scale(current at rest, with ambulation, worst & least in last 24 hours). The Numeric Rating Scale is a simple, widely used tool for measuring pain intensity. It consists of a 0-10 point scale. This will be measured after surgery in the PACU.
Numeric Rating Scale @POD14, @week 6, @week 12 - average pain, worst & least: last 7 days; current | From 14 days following surgery, 6 weeks from surgery and 12 weeks from surgery.
  Numeric Rating Scale measured at 14 days following surgery, then at 6 weeks following surgery and then 12 weeks following surgery. Measurements will range from average pain to worst pain to least amount of pain over the last 7 days and current pain.
Cumulative Opioid consumption (Oral morphine equivalents = OME): PACU, 0-24hours, 0 to 168 hours (7 days postoperatively) | from first time in PACU to 24hours after and then 168hours after
  Cumulative Opioid consumption (Oral morphine equivalents = OME): Post anesthesia care unit (PACU) at 0 and 24hours and 168 hours (i.e. 7 days postoperatively). The primary outcome is cumulative consumption in oral morphine equivalents starting from entry into the post-anesthesia care unit (PACU). This measure will be taken from EPIC via the MAR and documented in the study "MUD"; post-discharge, patient to report date/time of opioid use # of pills, dose in diary and documented in study "MUD". Measurements will be taken in PACU, 0-24hrs, 0-48 hrs and 0-168hrs following surgery.
Opioid-free patients through POD2 (0-48hrs), POD7 (0-168hrs), POD14 (0-day 14) | From start of trial to post operative day 2, 7 and 14
  Patients that no longer require opioid medications at Postoperative day 2 (48hrs), 7 (168hrs) and 14
Currently taking opioids & Opioid refills (Y/N, assessed @POD14, @6 week, @12 week) | From surgery to post operative day 14 week 6 and week 12
  If patient is currently taking opioids or getting Opioid prescription refills, answered as either yes or no and assessed on post operative day 14, at week 6 and week 12 following surgery.
Non-opioid analgesic use (POD0-48 hrs, 0-168 hrs) | From day of surgery to 48hours after and then 168hours after
  Analgesics used other than opioids on day of surgery, postoperative day 2 (i.e. 48 hrs) and day 7 (i.e. 168hrs)
Study medication discontinuation (% of patients who stopped the placebo/Suzetrigine day 0 through post-op day 7) | From surgery to the 7th day post operatively
  The percentage of patients who patients who stopped taking either the placebo drug or Suzetrigine within the first 7 days following surgery
Request for Suzetrigine refill after randomization period | From date if surgery till until end of study up to 2 years after surgery
  Number of patients that requested more or a refill of Suzetrigine after the randomization period was over
Patient satisfaction with pain management: @ POD2 and @POD7 | From date of surgery to 2 days following surgery and then again 7 days following surgery
  Patients will communicate there satisfaction with how well their pain is controlled this will be assessed 2 days and 7 days following surgery. Number on Scale out of 10 (where 0 is not satisfied, 10 is very satisfied)
Pain Interference: @ POD2 and @ POD7 | From date of surgery to post operative day 2 and 7
  Measuring how much since surgery Pain has interfered with normal day to day activities. This will be self reported using a number Scale (0-10, 0= no interference, 10= significant interference) on postoperative days 2 and 7. Patients will be asked; how much, since your surgery, has pain interfered with performing activities in bed such as turning, sitting up, and changing position? how much, since your surgery, has pain interfered with walking? how much, since your surgery, has pain interfered with your sleep? how much, since your surgery, has pain interfered with your mood?
HOOS, JR @ 6 weeks | Upto 30 days preoperatively to 6 weeks following surgery
  Hip dysfunction and Osteoarthritis Outcome Score for Joint Replacement (HOOS, JR) is a 0-100 scale that assesses hip pain and function, where a higher score indicates better hip health and a lower score indicates greater disability. This will be assessed preoperatively within 30 days of the surgery and then again 6 weeks post operatively. This measure will be extracted via EPIC or by a patient reported survey if not filled out in EPIC/mychart.
Incidence of adverse invents (POD0-7) | From the date the medication is given to the post operative day 7.
  Unexpected adverse events, that may occur to the patient after administration of Suzetrigine from the date the medication is given to the 7th day following surgery using Common Terminology Criteria for Adverse Events (CTCAE) v6.0 (MedDRA 28.0) grading system
  Grade 1 Mild; Grade 2 Moderate; Grade 3 Severe or medically significant; Grade 4 Life-threatening consequences; Grade 5 Death related to AE.
  for Nausea, Vomiting, Constipation, Difficulty passing urine, Concentrating, Somnolence, Lightheaded/dizziness, Confusion, Fatigue, Pruritis, Headache, Dry mouth, Paresthesia, Muscle spasm, Rashes, Problems with sleep, Delirium, Abnormal lab values, Other Patient-reported adverse effects (diarrhea, changes to heart beat/arrythmias, blurred vision, low blood pressure, difficulty breathing, hives, swelling of the face/lips/tongue/extremities/throat, other)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes